CLINICAL TRIAL: NCT01763658
Title: Evaluation of Oxidant Status in Patients With Immune Thrombocytopenia (ITP) and the Role of an Adjuvant Antioxidant Therapy
Brief Title: Oxidant Status and Effect of Antioxidant in Immune Thrombocytopenia
Acronym: ITP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohsen Saleh Elalfy, professor of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Antioxident in ITP
Record Dates: First submitted 2013-01-06; First posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP, antioxidant therapy, oxidant status
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Drug Therapy; Inosine Triphosphate; Dexamethasone; Prednisolone; Methylprednisolone Hemisuccinate; RHO(D) antibody; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antioxidant, drug therapy for ITP (Experimental): interventional arm 1 and will receive antioxidant therapy (Antox tablets ( 1 tablet contains : Vit. A 2000 IU, Vit C 90 mg, Vit E 15 mg and selenium yeast 55 ug ) with the therapy selected for ITP tailored according to patient's presentation.For Antox tablets it will be given daily for 6 months.
  Interventions: Drug: Antox tablets(Mepaco); Other: drug therapy for ITP
- drug therapy for ITP (Active Comparator): drug therapy for ITP according to ASH, 2011 guidelines.
  Interventions: Other: drug therapy for ITP

INTERVENTIONS:
Drug: Antox tablets(Mepaco) — effect of antioxidant on disease outcome
  Other Names: antioxidant drug
  Arms: Antioxidant, drug therapy for ITP
Other: drug therapy for ITP — drugs will be selected according to ASH,2011 guidelines
  Other Names: dexamethasone; prednisolone; solumedrol; Anti-D; intravenous immunoglobulin; romioplastin

SUMMARY:
Oxidative stress occurs as a result of increased activity of free radical-producing enzymes, decreased activity of free radical-removing enzymes, and insufficient levels of antioxidants. The most sensitive molecules to oxidation are lipids. Loss of cell membrane elasticity, increased cell fragility, and a shortened cellular life span results from oxidation of cell membrane lipids.

DETAILED DESCRIPTION:
Free oxygen radicals may have an effect on the structural and functional damage of platelets and plays a role in pathogenesis of thrombocytopenia in both, acute and chronic ITP.

Selenium is an essential mineral found in small amounts in the body. It works as an antioxidant, especially when combined with other antioxidants as vitamin E , A and C. Antioxidants neutralize free radicals and may reduce or even help prevent some of the damage they cause.

aim of this study is to assess oxidant and antioxidant systems initially in patients with acute and chronic immune thrombocytopenia (ITP) and 6 months later.Another aim of the study is to evaluate effect of antioxidant therapy on bleeding score, platelet count and antioxidant status during 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1. All patients less than 18 years with primary ITP; at initial presentation with platelet count less than 40 x 109/L attended Ain Shams Hematology clinic Children hospital from January 2013 and followed-up for 6 months.

  2. For acute ITP, patients will be newly diagnosed (about one month within the diagnosis).

  3. For chronic (12-24 months) and persistent (3-12 months) ITP patients.

Exclusion Criteria:

1. Patients' platelet count more than 40 x 109/L.; or above 18 years
2. Patients with secondary cause for thrombocytopenia.
3. Patients with any there associated chronic illness affecting oxidant status

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
oxidant status in ITP | 6 month
  oxidant and antioxidant systems initially in patients with acute and chronic immune thrombocytopenia (ITP)

SECONDARY OUTCOMES:
antioxidant therapy | 6 months
  antioxidant therapy on bleeding score, platelet count and antioxidant status

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen S Elalfy, professor, Principal Investigator — Ain Shams University
Locations (1):
- hematology clinic ,pediatrics hospital, Ain Shams University hospital Cairo, Egypt, Cairo, Egypt